CLINICAL TRIAL: NCT02029664
Title: Gait Control of Stroke Patients Using Visual Feedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Manager, National Rehabilitation Center, Seoul, Korea
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: NRC-2013-04-037
Record Dates: First submitted 2013-12-28; First posted 2014-01-08 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Visual feedback distortion (Experimental): Visual distortion increment based on the gait pattern
  Interventions: Device: Visual distortion increment based on the gait pattern

INTERVENTIONS:
Device: Visual distortion increment based on the gait pattern

SUMMARY:
The purpose of this study is to determine the possibility of gait pattern change via visual feedback among patients with stroke. Also, the optimal visual feedback would be chosen from this study.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke patients >= 18 years old
* Functional Ambulation Category >=3
* Cognitively intact enough to follow the study protocol
* Adults without any gait problem

Exclusion Criteria:

* Quadriplegic stroke patients
* Orthopedic problems to affect gait
* Underlying other neurological or psychological disorders
* Spasticity or contracture which impede the gait.
* Uncontrolled medical problems
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Step length symmetry | Participants will be followed for the duration of treadmill gait, an expected average of 15 minutes
  Step length symmetry during treadmill gait. When the participants walk on the treadmill, the walk symmetry was calculated from the sensor attached to them.
  During the whole period of treadmill gait, step length asymmetry will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, Seoul, South Korea

REFERENCES:
- See also: Related Info — http://www.nrc.go.kr/